CLINICAL TRIAL: NCT04902833
Title: Characterization Of Acquired Pyruvate Kinase Deficiency In Clonal Myeloid Neoplasms
Brief Title: Acquired Pyruvate Kinase Deficiency In Clonal Myeloid Neoplasms
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Hanny Al-Samkari, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 21-187
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pyruvate Kinase Deficiency; Pyruvate Kinase Deficiency Anemia; Hereditary Hemolytic Anemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm; Clonal Myeloid Neoplasm; Myeloproliferative Neoplasm; Acute Myeloid Leukemia; Clonal Cytopenia of Undetermined Significance; Other Clonal Myeloid Neoplasm; Unexplained Coombs-negative Non-immune Hemolytic Anemia
Keywords: Pyruvate Kinase Deficiency; Pyruvate Kinase Deficiency Anemia; Hereditary Hemolytic Anemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm; Clonal myeloid neoplasm; Myeloproliferative Neoplasm; Acute Myeloid Leukemia; Clonal Cytopenia of Undetermined Significance; Other clonal myeloid neoplasm; Unexplained Coombs-negative non-immune hemolytic anemia
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic, Congenital; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders; Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort I: Approximately 75 anemic (Hgb <11.0 g/dL) MDS Participants without overt clinical evidence of hemolysis.
  - Single Blood Draw
  Interventions: Procedure: Blood Draw
- Cohort 2: 25 Participants with clonal myeloid disorders of any type with evidence of non-immune, otherwise unexplained hemolytic anemia
  -Single Blood Draw
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Blood specimen 2-4 teaspoons

SUMMARY:
This cross-sectional prevalence assessment study involves a single blood draw in specific patient populations to assess for enzymatic and genomic evidence for acquired pyruvate kinase deficiency.

DETAILED DESCRIPTION:
This cross-sectional prevalence assessment study involves a single blood draw in specific patient populations to assess for enzymatic and genomic evidence for acquired pyruvate kinase deficiency.

* Red cell pyruvate kinase enzyme activity and next-generation sequencing (NGS) hereditary hemolytic anemia panels will be performed on samples from all recruited participants.
* The study will recruit patients to two separate cohorts.

  * Cohort 1 will recruit approximately 75 anemic (Hgb <11.0 g/dL) MDS participants without overt clinical evidence of hemolysis.
  * Cohort 2 will recruit approximately 25 participants with clonal myeloid disorders of any type with evidence of non-immune, otherwise unexplained hemolytic anemia
* Participation in the study involves a single blood draw. Basic information about the participant's blood disorder will also be collected.

It is expected that about 100 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1

  * Capable and willing to provide informed consent for participation in the study.
  * Diagnosis of clonal cytopenia of undetermined significance (CCUS), myelodysplastic syndrome (MDS) or myelodysplastic/myeloproliferative neoplasm (MDS/MPN syndrome) according to 2016 World Health Organization (WHO) classification system.
  * Anemia secondary to underlying clonal cytopenia of undetermined significance (CCUS), MDS or MDS/MPN syndrome, defined as a hemoglobin <11.0 g/dL measured within 30 days of study enrollment. Anemia should not be related to nutritional deficiency (such as iron, cobalamin, folate, or copper deficiencies), peripheral immune or non-immune hemolysis, or renal disease, in the opinion of the investigator.
  * Age >18 years.
* Cohort 2

  * Capable and willing to provide informed consent for participation in the study.
  * Diagnosis of a clonal myeloid neoplasm, such as MDS, MDS/MPN syndrome, myeloproliferative neoplasm (MPN), acute myeloid leukemia (AML), clonal cytopenia of undetermined significance (CCUS), or other clonal myeloid neoplasm according to 2016 World Health Organization (WHO) classification system.
  * A diagnosis of an otherwise unexplained Coombs-negative non-immune hemolytic anemia, according to the clinical judgement of the investigator. Some form of objective laboratory evidence must be present, including one or more of the following: negative direct antiglobulin (Coombs) test, reduced haptoglobin, elevated indirect bilirubin, elevated lactate dehydrogenase, elevated aspartate aminotransferase, or compatible findings on peripheral blood film. Results of all of these tests are not required to satisfy this criterion.
  * Age >18 years.

Exclusion Criteria:

* Cohort 1

  * Receipt of red cell transfusion within 60 days of study enrollment.
  * Have a known untreated nutritional anemia or acquired disorder resulting in hemolysis, such as paroxysmal nocturnal hemoglobinuria (PNH). A known hereditary anemia (such as thalassemia trait) is not exclusionary if the patient's baseline hemoglobin has worsened significantly (in the opinion of the investigator) after development and diagnosis of MDS.
* Cohort 2

  * Have a known hereditary anemic disorder, such as thalassemia, sickle cell disease, or hereditary enzyme deficiency, with the exception of hereditary X-linked glucose-6-phosphate dehydrogenase deficiency known not to cause chronic baseline hemolysis. Testing for these diagnoses is not required unless deemed clinically necessary.
  * Have a known untreated nutritional anemia or acquired disorder resulting in hemolysis, such as paroxysmal nocturnal hemoglobinuria (PNH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1 will recruit approximately 50 anemic (Hgb <11.0 g/dL) MDS patients without overt clinical evidence of hemolysis. Cohort 2 will recruit approximately 50 patients with clonal myeloid disorders of any type with evidence of non-immune, otherwise unexplained hemolytic anemia.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall prevalence of possible or likely acquired pyruvate kinase deficiency | Day 1
  defined by PK enzyme activity or PK:HK ratio >1 SD below the control mean (healthy subject mean) as measured by enzyme assay, or potentially pathogenic mutations in the PKLR gene as found on PKLR sequencing

SECONDARY OUTCOMES:
Overall prevalence of definite acquired pyruvate kinase deficiency | Day 1
  Defined by PK enzyme activity below normal (or a PK:HK ratio <8.7) as measured by enzyme assay, or known pathogenic mutations in the PKLR gene as found on PKLR sequencing
Red cell pyruvate kinase enzyme activity | 60 days
  Red cell pyruvate kinase enzyme activity in patients not receiving red cell transfusion in the 60 days prior to blood draw
Red cell pyruvate kinase | 60 Day
  hexokinase enzyme activity ratio in patients not receiving red cell transfusion in the 60 days prior to blood draw
Somatic mutations in PKLR (and other genes associated with acquired PKD) detected in the hematopoietic clone | Day 1
Somatic mutations in other genes associated with hemolytic anemia detected in the hematopoietic clone | Day 1
Characterization of pyruvate kinase-related red cell metabolites (ATP, 2,3-DPG) and pyruvate kinase-R protein in patients with clonal myeloid disorders | Day 1
Impact of pyruvate kinase activators on PK activity in vitro | Day 1

OTHER OUTCOMES:
Characterization of other possible factors involved in acquired PKD, including acquired epigenetic or gene expression factors | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Hanny Al-Samkari, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation